CLINICAL TRIAL: NCT06769607
Title: Evaluation of a Novel Auto-Adjusting Positive Airway Pressure Algorithm for the Treatment of Obstructive Sleep Apnea Clinical Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ResMed (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: SLP-24-10-01
Record Dates: First submitted 2024-11-11; First posted 2025-01-10 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Intervention Model Description: This is a blind, randomized cross over (or single arm) study aiming to show that the new algorithm is efficacious in the treatment of OSA. Furthermore, it allows for the comparison of relevant objective data parameters from the device, wearable data and subjective outcomes in comparison to an established algorithm.
  The study is planned in two phases. Phases may be repeated until sufficient confidence is gained of the intended behavior of the investigational algorithm and to ensure that the sample has appropriate coverage of different user experiences which can impact study outcomes (e.g. comfort settings such as soft response).
  After the conclusion of phase 1 and 2, participants who indicate that the experience on the investigational device was satisfactory and would like to continue using the algorithm will be included in an optional extended trial period.
Who Masked: Participant
Masking Description: Single (Participant)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Investigational algorithm (Experimental): The participants will trial the investigational algorithm and the control algorithm in a randomized order. Each will be used for up to 4 weeks in the home environment in place of their own device/therapy. The study device will be set up to align with the majority of the participants current therapy settings.
  Interventions: Device: Investigational algorithm
- Control algorithm (Active Comparator): The participants will trial the investigational algorithm and the control algorithm in a randomized order. Each will be used for up to 4 weeks in the home environment in place of their own device/therapy. The study device will be set up to align with the majority of the participants current therapy settings.
  Interventions: Device: Control algorithm

INTERVENTIONS:
Device: Investigational algorithm — Investigational algorithm developed for the treatment of Obstructive Sleep Apnea.
  Arms: Investigational algorithm
Device: Control algorithm — Released algorithm intended for the treament of Obstructive Sleep Apnea
  Arms: Control algorithm

SUMMARY:
This study aims to assess the effectiveness of an investigational algorithm in the treatment of obstructive sleep apnea.

DETAILED DESCRIPTION:
This is a blind, randomized cross over (or single arm depending on phase) study aiming to show that the new algorithm is efficacious in the treatment of obstructive sleep apnea (OSA). Furthermore, it allows for the comparison of relevant objective data parameters from the device and subjective outcomes in comparison to an established algorithm.

This study is planned in two phases. Phase 1 aims to gain confidence that the algorithm is functioning as intended, and allow for minor modifications to be made to the software before proceeding to Phase 2.

Phase 2 aims to assess the performance of the algorithm in a broader range of participants to capture data and subjective feedback comparing the users experience between the new algorithm and the control algorithm.

After the conclusion of phase 1 and 2, an optional extended trial period will be offered to participants who indicate that the experience on the investigational device was satisfactory and would like to continue using the algorithm will be included in an optional extended trial period.

The study will be conducted in the home environment. Participants who met the inclusion/exclusion criteria will be contacted. Participants will be explained the details of the trial and those who wish to take part will be invited to a selected site for the first study visit. In addition, subjects may be asked if they are willing to wear a wearable during both day and night (unless charging) for the duration of the study iteration. The wearable will be a commercially available wellness wearable that collects data to provide information about sleep and activity.

Visit 1 Participants will provide written informed consent. Participants will be set up on the algorithm they are first randomized to. If the participant and assessor are happy to proceed, the participants will take the device home to trial the first randomized algorithm, participants will be asked to complete a questionnaire regarding their therapy experience.

Visit 2 Participants will then be switched to the alternative algorithm and take the study device home to test. After trialling the second algorithm, participants will be asked to complete a questionnaire regarding their therapy experience and overall preferences.

Note: Visit 2 is not required if a cross over is not required in Phase 1.

Visit 3 The participant will return the investigational device to the assessor. The participants' questionnaire responses will be reviewed. Participants will be reimbursed. This concludes the participation in the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants willing to give written informed consent.
* Participants who can read and comprehend English.
* Participants who ≥ 18 years of age
* Participants who have been using a ResMed AirSense 10 or 11 device.
* Participants currently using AutoSet (APAP) mode.
* Participants being established on PAP therapy for the treatment of OSA for approximately >3 months.
* Participants who can participate in the study for up to 8 weeks.

Exclusion Criteria:

* Participants using Bilevel flow generators.
* Participants using CPAP, AutoSet for Her
* Participants who are or may be pregnant.
* Participants with a preexisting lung disease/ condition that would predispose them to pneumothorax (for example: COPD, lung cancer; fibrosis of the lungs; recent (< 2years) case of pneumonia or lung infection; lung injury.
* Participants believed to be unsuitable for inclusion by the researcher.
* Participants who are currently enrolled in other medical clinical studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-04-10 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Comparison of the algorithm efficacy (AHI) to a clinically relevant data | 8 weeks
  The mean residual AHI of the investigational algorithm will be compared against an excepted clinical benchmark of 5 using a one sample t test.

SECONDARY OUTCOMES:
Secondary endpoint: Device usage | From enrolment to the end of each study arm (up to 8 weeks)
  Hypothesis: the investigational algorithm will be equivalent or better than the comparison algorithm.
  Objective statistics on "Device usage" in hours per day (Hrs) stored in the PAP device will be downloaded. These parameters will be captured from each arm of testing and results will be analysed and compared.
Secondary endpoint: Leak | From enrollment to the end of each study arm (up to 8 weeks)
  Hypothesis: the investigational algorithm will be equivalent or better than the comparison algorithm.
  Objective statistics on "Leak" in litres per minute (L/min) stored in the PAP device will be downloaded. These parameters will be captured from each arm of testing and results will be analysed and compared.
Secondary endpoint: Pressure | From enrolment to the end of each study arm (up to 8 weeks)
  Hypothesis: the investigational algorithm will be equivalent or better than the comparison algorithm.
  Objective statistics on "Pressure" in centimeters of water (cmH2O) stored in the PAP device will be downloaded. These parameters will be captured from each arm of testing and results will be analysed and compared.
Secondary endpoint: Subjective scores | From enrolment to the end of each study arm (up to 8 weeks)
  Hypothesis: the investigational algorithm will be equivalent or better than the comparison algorithm and/or Criterion score of 6.
  Subjective scores will be collected from participants on each item (e.g. comfort, breathign comfort, ease of falling asleep). Scores will be collected using an 11-point Likert Scale where a score of 10 is considered very favorable whereas score of 0 is considered very unfavorable.
Wearable data - Sleep metrics | From enrolment to the end of each study arm (up to 8 weeks)
  Hypothesis: the investigational algorithm will be equivalent or better than the comparison algorithm. Objective statistics on sleep metrics measured via the wearable will be downloaded. These parameters will be captured from each arm of testing and results will be analysed and compared.
Wearable data - Activity Metrics | From enrolment to the end of each study arm (up to 8 weeks)
  Hypothesis: the investigational algorithm will be equivalent or better than the comparison algorithm. Objective statistics on activity metrics measured via the wearable will be downloaded. These parameters will be captured from each arm of testing and results will be analysed and compared.

CONTACTS AND LOCATIONS:
Locations (1):
- ResMed Ltd, Bella Vista, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No